CLINICAL TRIAL: NCT07300033
Title: Bioequivalence of Liquid Metformin (100 mg/mL and 250 mg/mL) and Immediate-Release Metformin Tablets: A Randomized, Crossover Study in Adult Subjects
Brief Title: Bioequivalence Study of Liquid Metformin (100 and 250 mg/mL) vs IR Tablets
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASP-018-Met
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Arm Crossover (Experimental)
  Interventions: Drug: Liquid Metformin 100 mg/mL; Drug: Liquid Metformin 250 mg/mL; Drug: Metformin Immediate-Release Tablet

INTERVENTIONS:
Drug: Liquid Metformin 100 mg/mL — A single oral dose of a liquid metformin formulation at a concentration of 100 mg/mL will be administered under fasting conditions in one treatment period of the crossover.
Drug: Liquid Metformin 250 mg/mL — A single oral dose of a liquid metformin formulation at a concentration of 250 mg/mL will be administered under fasting conditions in one treatment period of the crossover.
Drug: Metformin Immediate-Release Tablet — A single oral dose of standard immediate-release metformin tablet(s) will be administered under fasting conditions in one treatment period of the crossover.

SUMMARY:
This is an open-label, randomized, two-treatment, two-period crossover study evaluating the bioequivalence of liquid metformin formulations at 100 mg/mL and 250 mg/mL compared with immediate-release metformin tablets in healthy adult subjects. Each participant will receive both treatments in randomized sequence with an adequate washout interval between periods. Serial blood samples will be collected to assess metformin pharmacokinetics, and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 to 55 years of age, inclusive.

Body mass index (BMI) between 18.0 and 30.0 kg/m², inclusive.

Medically healthy based on medical history, physical examination, vital signs, clinical laboratory tests, and 12-lead ECG, in the opinion of the investigator.

Non-smoker or light smoker (10 or fewer cigarettes per day or equivalent) willing to abstain from smoking during confinement periods.

Able to understand and provide written informed consent prior to participation in the study.

Willing and able to comply with all study requirements, including fasting requirements and pharmacokinetic blood sampling.

Females of childbearing potential must use an acceptable method of contraception as determined by the investigator.

Exclusion Criteria:

* Known hypersensitivity or contraindication to metformin or any component of the study formulations.

History or presence of any clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic, or psychiatric disorder that, in the opinion of the investigator, could interfere with study participation or interpretation of results.

Estimated glomerular filtration rate (eGFR) less than 90 mL/min/1.73 m², or any clinically significant abnormal clinical laboratory findings.

History of lactic acidosis.

Use of prescription or over-the-counter medications, herbal supplements, or dietary supplements within 14 days before the first study dose, unless approved by the investigator.

Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV.

Positive urine drug screen or positive alcohol breath test at screening or admission.

Participation in another clinical trial or receipt of an investigational product within 30 days or 5 half-lives (whichever is longer) before the first study dose.

Donation of 450 mL or more of blood, or significant blood loss, within 8 weeks before first study dose.

Pregnant or breastfeeding females.

Women of childbearing potential not using acceptable contraception.

Any condition or situation that, in the opinion of the investigator, would make the participant unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC₀-t) of Metformin | Up to approximately 24 to 36 hours postdose in each treatment period
Maximum Observed Plasma Concentration (Cmax) of Metformin | Up to approximately 24 to 36 hours postdose in each treatment period

IPD SHARING:
Plan to Share IPD: No